CLINICAL TRIAL: NCT01674699
Title: Berlin Heart EXCOR Pediatric Post Approval Study
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Berlin Heart, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: EXCOR PAS; H100004 (Other: FDA)
Record Dates: First submitted 2012-08-27; First posted 2012-08-29 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2012-08

CONDITIONS: Severe Isolated Left Ventricular Dysfunction; Severe Biventricular Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- EXCOR: Pediatric candidates age 0 - 21 with severe isolated left ventricular or biventricular dysfunction who are candidates for cardiac transplant and require circulatory support may be treated using the EXCOR® Pediatric.
  Interventions: Device: EXCOR Pediatric

INTERVENTIONS:
Device: EXCOR Pediatric — Ventricular Assist Device
  Other Names: EXCOR Pediatric VAD; EXCOR Pediatric Ventricular Assist Device; Berlin Heart EXCOR Pediatric

SUMMARY:
The purpose of this post-approval study of the EXCOR® Pediatric VAD is to evaluate whether safety and outcomes of the device use in the commercial setting are comparable to the safety and outcomes of the device use in the IDE study.

DETAILED DESCRIPTION:
EXCOR® Pediatric is intended to provide mechanical circulatory support as a bridge to cardiac transplantation for pediatric patients. Pediatric candidates with severe isolated left ventricular or biventricular dysfunction who are candidates for cardiac transplant and require circulatory support may be treated using the EXCOR® Pediatric.

Study Purpose The purpose of this post-approval study of the EXCOR® Pediatric VAD is to evaluate whether safety and outcomes of the device use in the commercial setting are comparable to the safety and outcomes of the device use in the IDE study. Because the device had extensive use (available to all North American sites who requested the device under compassionate use regulations), it is expected that the pre-approval and post-approval use will be similar.

The primary safety objective of the EXCOR® Pediatric VAD Post-Approval Study is to demonstrate that the serious adverse event (SAE) rate in subjects implanted with the EXCOR® Pediatric in the study is not greater than the rate experienced in the IDE study.

The primary effectiveness objective for the EXCOR® Pediatric VAD Post Approval Study is to assess the outcome following implantation of the EXCOR® Pediatric for transplant eligible children in need of mechanical circulatory support. Outcome is defined as transplant, recovery of left ventricular function or death.

The following secondary objectives will be summarized:

* Device Malfunction
* Site evaluation of explanted pumps for suspected thrombus
* Assessment of the learning curve

The study will be an "all-comers" prospective study maintained by the sponsor consisting of pediatric patients aged 0-21 years implanted according to the IFU with the EXCOR® Pediatric who are transplant eligible children in need of mechanical circulatory support and who consent to be enrolled into the study.

The study will enroll at least 39 subjects implanted with the device per device labeling and who consent to be enrolled into the post approval study after the study commencement at any implanting site with IRB approval for participation.

Study enrollment is expected to take 10-12 months and subjects will be followed until they reach an outcome. The primary endpoints will be analyzed and reported to FDA during the regular reporting cycle. Explanted subjects will be followed for 24 months post explant. A final report will be submitted to FDA once all subjects complete their 24 month post explant visit. Average time on device is expected to be similar to the average time on the device during the IDE study (58 days) therefore the last implant is expected to be followed until outcome (IDE range was 0 - 435 days). The overall study duration is expected to be approximately 36-38 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient requires mechanical circulatory support and is eligible for cardiac transplantation
* Legal guardian and patient (if age appropriate) understands the nature of the implant procedure and are willing to comply with associated follow-up evaluations, and provide written informed consent and assent prior to the procedure

Exclusion Criteria:

* Patient is currently enrolled in EXCOR® Pediatric pre-market study
* Patient is currently participating in another investigational device or drug trial which would confound the results of the study

Ages: 1 Day to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study will be an "all-comers" prospective study including subjects whom meet the Inclusion and Exclusion Criteria. Pediatric candidates with severe isolated left ventricular or biventricular dysfunction who are candidates for cardiac transplant and require circulatory support may be treated using the EXCOR® Pediatric.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Estimated)
Dates: Start 2012-08; Primary Completion 2015-06 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Safety | 2 years
  The primary safety objective of the EXCOR® Pediatric VAD Post-Approval Study is to demonstrate that the serious adverse event (SAE) rate in subjects implanted with the EXCOR® Pediatric in the study is not greater than the rate experienced in the IDE study.
Effectiveness | 2 years
  The primary effectiveness objective for the EXCOR® Pediatric VAD Post Approval Study is to assess the outcome following implantation of the EXCOR® Pediatric for transplant eligible children in need of mechanical circulatory support. Outcome is defined as transplant, recovery of left ventricular function or death.

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Kroslowitz, BS, Study Director — Berlin Heart, Inc